CLINICAL TRIAL: NCT00275600
Title: Randomized Clinical Trial of Vitamin E and Evening Oil of Primrose for the Managment of Cyclical Breast Pain
Brief Title: Randomized Clinical Trial of Vitamin E and Evening Oil of Primrose for the Managment of Breast Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: New Health International (Unknown)
Responsible Party: Sandhya Pruthi, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1957-02
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2009-11

CONDITIONS: Cyclical Breast Pain
MeSH Terms: interventions — Vitamin E

INTERVENTIONS:
Drug: Vitamin E, Evening Oil of Primrose, and Placebo

SUMMARY:
This study is being done to find out what effects Vitamin E or Evening Oil of Primrose has on cyclical breast pain.

DETAILED DESCRIPTION:
Cyclical mastalgia is a common complaint of women presenting to their primary care physicians. Cyclical breast pain is defined as prementstrual breast discomfort associated with hormonal fluctuations during the menstrual cycle. A clinical breast examination and sometimes additional imaging, such as sonography or mammography, is required as part of the evaluation to exclude malignancy. For most women, the symptoms are effectively managed with reassurance and conservative treatment measures such as the use of a supportive bra or over the counter pain medication such as acetaminophen or anti-inflammatories. However, a small number of women will require additional drug treatment with danazol after failing to respond to conservative measures. Unfortunately, danazol is associated with significant side effects. In the Mayo Breast Clinic, women with cyclical breast pain are managed with Vitamin E and Evening oil of primrose (EOP) either as single agents or in combination. These over the counter supplements are readily available, acceptable due to minial side effects and appear to lead to significant reduction in breast pain. We propose a randomized placebo controlled trial to determine if any vitamin E or EOP or the combination of both are effective in managing cyclical breast pain.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* premenopausal
* cyclical breast pain
* breast pain survey indicating 3 or more on scale of 1-10
* if > 40 years of age, need normal mammogram and/or ultrasound if indicated and if not done within the last year
* if < 40 years of age, a directed ultrasound in the area of pain
* can be on oral contraceptives

Ages: 18 Years to 56 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2003-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Test if Vitamin E improves cyclical breast pain
Test if Evening Oil of Primrose improves cyclical breast pain
Test if combination of Evening Oil of Primrose and Vitamin E works synergistically for cyclial breast pain

CONTACTS AND LOCATIONS:
Overall Officials: Sandhya Pruthi, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States